CLINICAL TRIAL: NCT00255229
Title: Study of Glutamine as Prophylaxis for Irinotecan Induced Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GI-05-0024
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: irinotecan; 5FU; amino acids; heat shock protein
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Irinotecan, 5FU, Glutamine
  Interventions: Drug: Glutamine
- 2 (Placebo Comparator): Irinotecan, 5FU, Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glutamine — Glutamine 10 g four times daily starting two days before treatment for six days in total
  Arms: 1
Other: Placebo — Glutamine placebo
  Arms: 2

SUMMARY:
Irinotecan (7-ethyl-10- {4(-1-piperidino)-1-piperidino} carbonyloxy camptothecin) is a semisynthetic camptothecin derivative introduced in the 1980's. Irinotecan is a prodrug metabolized by carboxylesterases to an active metabolite 7-ethyl-10-hydroxy-camptothecin (SN38). SN38 exerts its cytotoxic effect by forming stable complexes with topoisomerase I and DNA. These complexes collide with replication forks and cause breaks in DNA. Studies substantiated irinotecan's activity in 5FU resistant colorectal cancer and led to its approval for treatment of 5FU resistant colorectal cancer in the United States, Canada and Europe.Colorectal cancer studies demonstrated that single agent irinotecan's dose limiting toxicity was diarrhea occurring 5 to 6 days after its administration. High dose loperamide at first occurrence of diarrhea has decreased the incidence of diarrhea but the incidence of grade 3/4 diarrhea remains high at 28 to 40%.

ELIGIBILITY:
Inclusion Criteria:

* metastatic colorectal cancer to be treated with FOLFIAT chemo

Exclusion Criteria:

* severely abnormal liver and kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Reduction in diarrhea. | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada